CLINICAL TRIAL: NCT06461013
Title: The Effect of Blood Flow Restriction Training on Lower Limb Motor Function in Stroke Patients With Hemiplegia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sorry, the treatment protocol has been changed. Withdrawn: Study halted prematurely, prior to enrollment of first participant
Sponsor: Yunhong Tian (Other Government)
Responsible Party: Sponsor-Investigator, Yunhong Tian, Principal Investigator, Nanchong Central Hospital
Organization: Nanchong Central Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023ER378-1
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Hemiplegia and/or Hemiparesis Following Stroke
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine rehabilitation (No Intervention): Bridge exercise: Before conducting specific tests, participants should familiarize themselves with the relevant test actions and procedures. The key points of bridge exercise are: the subject is placed in a supine position, with both hands crossed in the center of the abdomen, the knee joint flexed, both feet flat on the bed surface, and the buttocks lifted off the bed surface with force. The patient is instructed to do bridge exercise as much as possible until the knee joint, hip joint, and neck are on the same line, which is considered qualified for bridge exercise;
- routine rehabilitation+blood flow restriction training (Experimental): Bridge exercise: Before conducting specific tests, participants should familiarize themselves with the relevant test actions and procedures. The key points of bridge exercise are: the subject is placed in a supine position, with both hands crossed in the center of the abdomen, the knee joint flexed, both feet flat on the bed surface, and the buttocks lifted off the bed surface with force. The patient is instructed to do bridge exercise as much as possible until the knee joint, hip joint, and neck are on the same line, which is considered qualified for bridge exercise;
  Interventions: Behavioral: Blood flow restriction

INTERVENTIONS:
Behavioral: Blood flow restriction — A common clinical tourniquet (7cm * 50cm in size) is placed in the middle section of the patient's thigh on the affected side, connected to a pressure gauge, observed and gradually pressurized to 160-170mmHg for about 10 minutes, then depressurized for 1 minute, and then re pressurized to 160-170mmHg. Each training session lasts for 20 minutes, once a day, five times a week, for a total of 8 weeks.
  Arms: routine rehabilitation+blood flow restriction training

SUMMARY:
flow restriction training combined with routine rehabilitation training can promote the recovery of lower limb muscle strength on the hemiplegic side of stroke patients, improve the lower limb motor function of patients, and further improve their daily life and walking ability. It provides a new treatment method for stroke patients with hemiplegia that leads to lower limb function loss and activity disorder, and the therapy also has the advantages of simple operation, high safety, good patient compliance and low cost, which is worthy of further clinical research and promotion.

DETAILED DESCRIPTION:
In this work, Stroke is a disease with a high incidence, high mortality and high disability rate, and it is becoming increasingly common in young individuals. More than 50% of these patients have long-term chronic motor dysfunction due to unilateral limb dysfunction, and abnormal limb movement patterns occur due to unilateral limb weakness, abnormal muscle tone and other symptoms, which can manifest as a typical "hemiplegic gait" on walking. Motor dysfunction after stroke, including muscle strength, dystonia and abnormal gait, is the main dysfunction, which can cause cardiopulmonary function decline, thrombosis, muscle atrophy, etc., reducing the ability of daily living and quality of life of patients. Routine rehabilitation training methods for stroke patients with dysfunction include muscle strength training techniques, neurodevelopmental treatment (NDT), motor relearning programs (MRPs), constraint-induced movement therapy (CIMT), neuromuscular electrical stimulation (NMES). But it cannot achieve a good rehabilitation treatment effect. Therefore, we found through lower extremity motor function (LE-FMA), balance function (BBS), activities of daily living (MBI), patients' walking distance (6-MWT test) and the MMT assessment of muscle strength of iliopsoas, quadriceps, hamstrings and tibialis anterior muscles testing that combining blood flow restriction training on the basis of traditional rehabilitation is beneficial for patient muscle rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of stroke meets the diagnostic criteria revised by the Fourth National
* Conference on Cerebrovascular Diseases
* Confirmed by cranial CT and/or MRI
* First onset, hemiplegia of one limb, clear consciousness, stable vital signs, no serious complications such as heart, lung, kidney, etc., no serious cognitive or audio-visual impairment

Exclusion Criteria:

* Uncontrolled hypertension
* Coronary artery disease
* Uncontrolled autonomic reflex abnormalities
* Severe spasms
* History of fractures or fractures
* Deep vein thrombosis
* Cognitive impairment, inability to cooperate

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Lower extremity subscale of Fugl-Meyer motor function assessment (LE-FMA) | 5 times a week for 8 weeks.
  The total score of lower limb motor function is 34 points, including 7 major items and 17 minor items. Each minor item has three score levels of 0, 1 and 2. Zero points means that the action cannot be performed, 1 point means that the action can only be partially completed, and 2 points means that the action can be fully completed. The higher the score, the better the lower limb motor function of patients. This scale is widely used in the rehabilitation evaluation of hemiplegic patients and can reflect the lower limb motor function of patients.
Berg Balance Scale (BBS) | 5 times a week for 8 weeks.
  The total score of the scale was 56 points, and there were 14 test items. Each item was rated from 0 to 4. A score of 4 indicated that the patient could perform the needed actions well, and a score of 0 indicated that the patient could not perform the actions at all. The higher the score is, the better the balance ability of the patient.
The Modified Barthel Index (MBI) | 5 times a week for 8 weeks.
  used to evaluate the ability of patients to perform activities of daily living, including the ability to complete daily tasks such as eating, moving, dressing, and walking. The higher the score is, the better the function. The activities related to lower limb function selected in this study included walking, moving, going upstairs, and toileting, with a total of 55 points.
6-Min Walking Test (6MWT) | 5 times a week for 8 weeks.
  The patient is asked to walk as far as possible along a 30-m minimally trafficked corridor for a period of 6 min, with the primary outcome measure being the 6-min walk distance measured in meters.
Manual muscle testing (MMT) | 5 times a week for 8 weeks.
  Muscle strength refers to the maximum force generated by muscle contraction, ranging from 0-5 grades from low to high. Freehand muscle strength measurement means that the examiner uses the freehand measurement method to make the patient move in different ways to eliminate the influence of compensation or borrowing force and measure the muscle strength of the target muscle group.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhangqin, Nanchong, Sichuan, China

IPD SHARING:
Plan to Share IPD: No